CLINICAL TRIAL: NCT03764969
Title: Modification of the Imbalance Between Goal-directed and Habitual Behavior in Human Addiction
Brief Title: Modification of Goal-directed and Habitual Behavior in Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRR265 C01
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use Disorder
Keywords: Addiction; Nicotine; Smoking Cessation; Relapse; Craving; habitual behavior; cognitive remediation; implicit priming; pavlovian instrumental transfer
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive; Smoking Cessation; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard smoking cessation program (SCP) (Active Comparator): standard smoking cessation program
  Interventions: Behavioral: standard smoking cessation program (SCP)
- SCP + CRT (Experimental): SCP plus cognitive remediation treatment (CRT)
  Interventions: Behavioral: standard smoking cessation program (SCP); Behavioral: Cognitive remediation treatment (CRT)
- SCP + ICHT (Experimental): SCP plus an implicit computer-based habit-modifying training (ICHT)
  Interventions: Behavioral: standard smoking cessation program (SCP); Behavioral: Implicit computer-based habit-modifying training (ICHT)

INTERVENTIONS:
Behavioral: standard smoking cessation program (SCP) — Each subject will receive standard SCP as group treatment once a week (1 hour) over six weeks. This group therapy is based on behavioural therapy and a psycho-educational approach (for more details see Batra & Buchkremer 2004), and will be carried out by a qualified therapist.
Behavioral: Cognitive remediation treatment (CRT) — Cognitive remediation treatment (CRT) employing a chess-based battery of tasks two times per week over six weeks as a group treatment in our outpatient clinic (60 min duration per session).
  Arms: SCP + CRT
Behavioral: Implicit computer-based habit-modifying training (ICHT) — Implicit computer-based habit-modifying training (ICHT), applied twice a week for six weeks. In this training, the participants perform a two-part training. First, a subliminal presentation (20 ms) of negative valenced primes before smoking-cues in context and secondly, a subliminal presentation of positive valenced primes before potentially reinforcing events.
  Arms: SCP + ICHT

SUMMARY:
This study aims to examine the modification of the hypothesized imbalance between goal-directed and habitual behavior and its neural correlates in smokers. Two interventions will be used as add-on trainings to a smoking cessation program.

DETAILED DESCRIPTION:
In this study, the investigators aim to assess the imbalance between goal-directed and habitual behavior, its neural basis and how it can be differentially modified in treatment-seeking smokers, using two training interventions. The first intervention is cognitive remediation treatment (CRT), also known as cognitive enhancement therapy, focusing on improving inhibitory control and executive functions. The second intervention, a computer-based habit-modifying training focusing on implicit drug seeking ("implicit computer-based habit-modifying training", ICHT) uses a conditioning approach through implicit priming and contextual modulation. Indicators of the imbalance will be examined with respect to reward devaluation, cue reactivity and a pavlovian instrumental transfer (PIT) paradigm. The investigators hypothesize that both interventions change the balance between goal-directed and habitual behavior but by different mechanisms. Whereas CRT should directly increase cognitive control, in contrast, ICHT should affect the early processing and the emotional valence of smoking and smoking cues.

ELIGIBILITY:
Inclusion Criteria:

* severe tobacco use disorder (TUD) according to DSM-5
* sufficient ability to communicate with investigators and answer questions in both written and verbal format
* ability to provide fully informed consent and to use self-rating scales

Exclusion Criteria:

* severe internal, neurological, and/or psychiatric comorbidities; other Axis I mental disorders other than TUD according to ICD-10 and DSM 5 (except for mild depression, i.e. F32.0, adjustment disorder and specific phobias) in the last 12 months
* history of brain injury
* severe physical diseases
* common exclusion criteria for MRI (e.g. metal, claustrophobia)
* positive drug screening (opioids, benzodiazepines, barbiturates, cocaine, amphetamines)
* psychotropic medication within the last 14 days
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Change in imbalance between goal-directed and habitual behavior | 2 time points: before and after 6 weeks SCP
  measured by reward devaluation procedure (Hogarth & Chase 2011)
Change in implicit smoking-related associations | 3 time points: before and after 6 weeks SCP plus after 3 months
  smoking-related implicit association task (Wiers et al. 2016).
Change in attentional bias to smoking cues | 3 time points: before and after 6 weeks SCP plus after 3 months
  smoking-related dot-probe task (Vollstädt-Klein et al. 2009).
Change in smoking urges | 3 time points: before and after 6 weeks SCP plus after 3 months
  questionnaire of smoking urges (QSU, Müller et al. 2001)); self-report questionnaire; two subscales: "intention and desire to smoke / anticipation of pleasure from smoking" (range 11 - 77) and "anticipation of relief from negative affect and nicotine withdrawal / urgent and overwhelming desire to smoke" (range 10 - 70) high values represent high craving
Change in working memory capacity | 3 time points: before and after 6 weeks SCP plus after 3 months
  Spatial Working Memory task from the Cambridge Automated Neuropsychological Test Automated Battery (Robbins et al. 1994)
Change in planning ability | 3 time points: before and after 6 weeks SCP plus after 3 months
  One Touch Stockings of Cambridge task from the Cambridge Automated Neuropsychological Test Automated Battery (Robbins et al. 1994)
Change in cognitive flexibility | 3 time points: before and after 6 weeks SCP plus after 3 months
  Internal-External Set Shifting task from the Cambridge Automated Neuropsychological Test Automated Battery (Robbins et al. 1994)

SECONDARY OUTCOMES:
nicotine consumption | 3 months follow-up
  self-report
Change in neural PIT effect | 2 time points: before and after 6 weeks SCP
  PIT phase of a choice task (adapted from Hogarth & Chase 2011)
Change in neural cue reactivity | 2 time points: before and after 6 weeks SCP
  fMRI cue-reactivity task (Vollstädt-Klein et al. 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim; Herta Flor, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Karl D, Wieland A, Shevchenko Y, Grundinger N, Machunze N, Gerhardt S, Flor H, Vollstadt-Klein S. Using computer-based habit versus chess-based cognitive remediation training as add-on therapy to modify the imbalance between habitual behavior and cognitive control in tobacco use disorder: protocol of a randomized controlled, fMRI study. BMC Psychol. 2023 Jan 25;11(1):24. doi: 10.1186/s40359-023-01055-z. PMID 36698210